CLINICAL TRIAL: NCT04005950
Title: Evaluation and Comparison of a Modified Skalpell-Bougie-technique for Cricothyreotomie: Comparison of a Conventional and a Realistic Self-modified Model
Brief Title: Comparison of a Conventional and a Realistic Self-modified Model
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Nina Pirlich, Dr. med., Principle Investigator, Johannes Gutenberg University Mainz
Other Study IDs: ScalpelCric Advanced
Record Dates: First submitted 2019-06-30; First posted 2019-07-02 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Cricothyroidotomy; Difficult Airway; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- medical doctors
  Interventions: Device: Scalpel Bougie technique; Device: modified Scalpel Bougie technique
- paramedics
  Interventions: Device: Scalpel Bougie technique; Device: modified Scalpel Bougie technique

INTERVENTIONS:
Device: Scalpel Bougie technique — ScalpelCric Set
Device: modified Scalpel Bougie technique — ScalpelCric Set plus speculum

SUMMARY:
According to the recently published german guidelines for the prehospital airway management regular training for cricothyroidotomy is recommended.

Even though participants prefer animal or cadaver trainingmodels, it is not possible to perform this comprehensive for a large number of participants due to organizational requirements like food hygiene, limited shelf-life and preparation time and expense.

Therefore the investigators modified an available for purchase cricothyroidotomy trainer (the AirSim Combo X) with everyday suitable and cost-effective utensils.

As a control group the investigators used a conventional simple plastic model.

DETAILED DESCRIPTION:
Obesity is an important risk factor for a cannot intubate cannot ventilate situation. Obese patients are more likely to require a cricothyroidotomy, due to failure rates of routine airway management. Relevant landmarks can be difficult to palpate. And the greater depth of the soft tissues overlying the larynx. Due to this reasons the investigators modified the adult intubation manikin AirSim Combo X with a drunk baby diaper to simulate the neck of an obese patient.

As a further modification the investigators prepared freezer bags filled with faked blood to simulate a possible bleeding.

35 medial doctors of the department of anesthesiology and 35 paramedics are going to perform two cricothyroidotomies in each model.

For the one time participants use the ScalpelCric Set and for the other time participants use the ScalpelCric Set plus a speculum.

Primary endpoint is the evaluation of reality of the two different manikins.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* german language in speaking and writing
* capability of giving consent

Exclusion Criteria:

* participants unwilling or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: medical doctors of the Department of anesthesiology of the University hospital Mainz, Germany
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2019-07-21 (Actual)

PRIMARY OUTCOMES:
evaluation of realistic applicability | 12 minutes
  using Likert scale (1=very realistic, 2= realistic, 3= not very realistic, 4=unrealistic)

SECONDARY OUTCOMES:
Time from initial handling equipment to a successful placement of the tracheal cannula | 300 seconds

OTHER OUTCOMES:
Number of trials | up to 12 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Johannes Gutenberg - Universität, Mainz, Rhineland-Palatinate, Germany